CLINICAL TRIAL: NCT06254196
Title: Randomized Clinical Trial of Telenursing for Monitoring Supportive Care Needs in Patients With Lung Cancer and Melanoma Candidates for the First Prescription of Targeted Therapies
Brief Title: Clinical Trial of Telenursing for Monitoring Supportive Care Needs in Patients With Lung Cancer and Melanoma Candidates for the First Prescription of Targeted Therapies
Acronym: Telenursing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RS1851/23
Record Dates: First submitted 2023-12-11; First posted 2024-02-12 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Lung Neoplasm; Melanoma
MeSH Terms: conditions — Lung Neoplasms; Melanoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: current clinical practice (No Intervention)
- Experimental group: Telenursing intervention (Experimental)
  Interventions: Procedure: Telenursing interventions for monitoring Supportive Care Needs

INTERVENTIONS:
Procedure: Telenursing interventions for monitoring Supportive Care Needs — Use of the Intelligence2health platform, data collection forms on Google Forms, and dedicated telephone line for telenursing remote nursing monitoring interventions.
  Based on the data, nurses will be able to implement patient education interventions aimed at preventing and monitoring healthcare support needs related to treatment.
  Arms: Experimental group: Telenursing intervention

SUMMARY:
Single-center, randomized clinical trial (RCT) with low intervention level (Telenursing), for the monitoring of patients affected by lung cancer and melanoma who are candidates for first prescription with Targeted Therapies. The study population will consist of patients suffering from lung cancer and melanoma. The objective of the study will be to evaluate the effectiveness of a Telenursing intervention, comparing the mean score of the total SCNs scale (Supportive Care Needs) after one month of treatment in the treatment arm and in the control arm.

Enrolled patients will then be randomized into two treatment arms:

* Arm 1 (Control Group): current clinical practice
* Arm 2 (Experimental group): Telenursing intervention.

DETAILED DESCRIPTION:
To cope with the welfare limits imposed from the SARS-CoV2 pandemic, the specialists of the I.R.C.C.S. Hospital Physiotherapy Institutes (IFO) of Rome have increased the use of telemedicine and have started teleassistance projects in various fields, especially in the nursing field.

The study: single-centre, randomized clinical trial (RCT) with a low level of intervention (Telenursing), for the monitoring of patients affected by lung cancer and melanoma who are candidates for first prescription with Targeted Therapies.

In particular:

Patients enrolled in arm 1 will follow clinical practice with in presence visits and paper based questionnaire and tools, filled daily and periodically (1, 3, 6 months)

Patients in arm 2 will use the Intelligence2health platform for telenursing interventions. For data collection, questionnaires on Google Forms will be used for the acquisition and control of data entered daily and periodically (1, 3, 6 months) by patients. A dedicated company telephone line for short communications will also be available to patients.

Through a greater nursing intervention, this clinical trial will assess the impact of a telenursing intervention on monitoring and improving the supportive care needs and the treatment experience of candidate patients to the first prescription of Targeted Therapies for lung cancer and melanoma.

The main objective is set to evaluate the effectiveness of a Telenursing intervention, choosing to compare the mean score of the total SCNs scale (Supportive Care Needs) after one month of treatment in the treatment arm and in the control arm.

Furthermore, among the secondary objectives we will evaluate Supportive Care Needs over time (until the end of the study after 6 months), the quality of life, the degree of patient satisfaction, the therapeutic adherence and finally the incidence and degree of severity of all Adverse Events (grade 1, 2, 3, 4 and 5 according to the Common, Terminology Criteria for Adverse Event, CTCAE).

The study will also explore the differences between the Adverse Events reported by healthcare personnel and those reported by patients (Patient Reported Outcomes, PROs), trying to develop a specific one nursing reporting system for the remote management of Adverse Events oncology.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 75;
* patients suffering from lung cancer and melanoma candidates for the first prescription with Targeted Therapies in exclusive treatment;
* patients able to understand, speak Italian and join the study by signing of paper informed consent;
* possibility of accessing and using the information technologies adopted in trial through a PC/tablet and personal internet connection;
* patients willing to comply with study procedures.

Exclusion Criteria:

* patients not suffering from lung cancer or melanoma;
* patients already treated or currently being treated with Targeted Therapies, or other treatment (chemotherapy and/or radiotherapy and/or exclusive palliative care);
* patients with cognitive problems, psychiatric disorders and poor compliance who could interfere with study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the nursing intervention. | 6 month
  Evaluate the effectiveness of the Telenursing nursing intervention by comparing the average score after one month of treatment on the total SCN (Supportive Care Needs) scale in the treatment arm and in the control arm, using the Supportive Care Needs monitoring form, to the measurement of adverse events using the 1-5 Likert scale - filled in by clinicians and by research nurses during the monthly in-person visit, according to the Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Need for supportive care | 6 months
  Assess the need for supportive care over time from the start of the trial to the end of the study.
Evaluate the incidence and severity of Adverse Events. | 6 months
  Evaluate the incidence and degree of severity of all Adverse Events in grades 1, 2, 3 and 4 according to the Common, Terminology Criteria for Adverse Event, CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Aurora De Leo, Nursing, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

REFERENCES:
- [Derived] De Leo A, Liquori G, Spano A, Panattoni N, Dionisi S, Iacorossi L, Giannetta N, Terrenato I, Di Simone E, Di Muzio M, Petrone F. Effect of Telenursing on Supportive Care Needs in Patients with Melanoma and Lung Cancer on Targeted Therapies: A Randomised Controlled Trial Study Protocol. Methods Protoc. 2024 Oct 3;7(5):78. doi: 10.3390/mps7050078. PMID 39452792